CLINICAL TRIAL: NCT06789978
Title: Prehospital Extracorporeal Cardiopulmonary Resuscitation: A Pilot Study in Prague
Brief Title: Rapid Prehospital ACcess to ECPR in Prague
Acronym: RACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Jan Bělohlávek, MD, PhD, professor, General University Hospital, Prague
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 134/23 S-IV
Record Dates: First submitted 2025-01-16; First posted 2025-01-23 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Out of Hospital Cardiac Arrest; Extracorporeal Cardiopulmonary Resuscitation
Keywords: Cardiac arrest; ECPR; ECMO; Prehospital
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Intervention Model Description: Single-arm interventional study with a historical control from Prague OHCA study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prehospital extracorporeal cardiopulmonary resuscitation (ECPR) (Experimental): Prehospital ECPR will include all patients who enter the study and receive ECPR.
  The historical control group will consist of patients from the Prague OHCA study who received in-hospital ECPR and fulfilled all relevant inclusion and exclusion criteria for this study.
  Interventions: Other: Extracorporeal cardiopulmonary resuscitation (ECPR)

INTERVENTIONS:
Other: Extracorporeal cardiopulmonary resuscitation (ECPR) — Prehospital extracorporeal cardiopulmonary resuscitation (ECPR)

SUMMARY:
A prospective pilot feasibility study of prehospital ECPR in patients with refractory OHCA

DETAILED DESCRIPTION:
The aim of this pilot prospective study is to assess the feasibility and effectiveness of a prehospital extracorporeal cardiopulmonary resuscitation (ECPR) system for refractory out-of-hospital cardiac arrest (OHCA) in Prague, compared to a historical cohort of in-hospital ECPR recipients from the Prague OHCA trial.

ELIGIBILITY:
Inclusion Criteria:

* Estimated age 18-70 years
* Refractory out-of-hospital cardiac arrest (3 unsuccessful defibrillations and/or at least 10 minutes of resuscitation in case of pulseless electrical activity)
* Witnessed cardiac arrest
* ECPR team available
* ECPR team alert within 20 minutes from the emergency call

Exclusion Criteria:

* Unwitnessed cardiac arrest
* Asystole
* ETCO2 less than 10 mmHg upon ECPR team arrival
* Known limitations of intensive care (Do Not Resuscitate - DNR status)
* Known severe neurological impairment prior to cardiac arrest (mRS 4-6)
* Suspected or known pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-06-16 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Time from collapse to ECPR | Time from estimated collapse to start of VA ECMO flow (estimated range: 20-100 minutes)
  Time from collapse to start of VA ECMO flow

SECONDARY OUTCOMES:
All cause survival at 30-days | 30-days
  Kaplan Meier analysis, log-rank test
Modified Rankin Scale at 30-days | 30-days
  Modified Rankin Scale (mRS) at 30 days: mRS 0-3 is considered a good outcome, and mRS 4-6 is considered a poor outcome.

OTHER OUTCOMES:
Major bleeding | 30-days
  Major bleeding, TIMI classification
Vascular complications | 30-days
  Vascular complications including disections, pseudoaneurysm, closure, thrombus
Infectious complications | 30-days
  Local groin infection requiring treatment or sepsis requiring treatment

CONTACTS AND LOCATIONS:
Locations (1):
- General University Hospital in Prague, Prague, Czechia, Czechia

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and analyzed in this study will be available from the principal investigators upon reasonable request.